CLINICAL TRIAL: NCT03828851
Title: Development of Domiciliary Program on Improving Activities of Daily Living Program for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201712067RIND
Record Dates: First submitted 2019-01-13; First posted 2019-02-04 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): ADL training program.
  Interventions: Other: Domiciliary care - Activities of Daily Living
- Control group (No Intervention): Receive rehabilitation program in the hospital.

INTERVENTIONS:
Other: Domiciliary care - Activities of Daily Living — Home-based ADL training.
  Arms: Experimental group

SUMMARY:
The purpose of this study was to investigate the effects of the Domiciliary care- Activities of Daily Living program on activities of daily living (ADL), motor, cognition, perception, sensory, quality of life, and depression for patients with stroke.

DETAILED DESCRIPTION:
Administering ADL and recovery of ADL functions are the primary efficacy indicators in long-term care and the main treatment goals in rehabilitation for patients with stroke. Residential rehabilitation is a direct way to observe patients' living environment and provides feasible ADL treatment plans for patients with stroke living at home or in the community. The purpose of this study was to investigate the effects of the Domiciliary care- Activities of Daily Living program on activities of daily living, motor, cognition, perception, sensory, quality of life, and depression. The eligible participants were recruited and assigned into two groups: ADL home program and control group who received traditional rehabilitation in hospital. The primary outcome measures were the Canadian Occupational Performance Measure, the Barthel Index-based Supplementary Scales, the Frenchay Activities Index, and ADL domain of the Stroke Impact Scale. The secondary outcome measures were the Fugl-Meyer Assessment, the Mini Mental State Examination, the Test of Visual Perceptual Skills-Third Edition, and the Center of Epidemiological Study-Depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Aged > 20 years
* Score 2-4 of the modified Rankin Scale
* Capability of following instructions
* Willing to participants to the study

Exclusion Criteria:

* Diagnoses of dementia and Parkinson's disease
* Physical limitations because of orthopedics diseases
* Peripheral nerve injury

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Changes of the Canadian Occupational Performance Measure | 6 months
  The Canadian Occupational Performance Measure assesses occupational performance. The total score ranges from 1-10. A higher score indicates better occupational performance. Changes of occupational performance will be assessed at the 6 weeks, 12 weeks, and 6 months.
Changes of the Barthel Index-based Supplementary Scales | 6 months
  The Barthel Index-based Supplementary Scales assesses basic activities of daily living. The total score range from 0-58. A higher score indicates better basic activities of daily living. Changes of basic activities of daily living will be assessed at the 6 weeks, 12 weeks, and 6 months.
Changes of the Frenchay Activities Index | 6 months
  The Frenchay Activities Index assesses instrumental activities of daily living. The total score range from 0-45. A higher score indicates better instrumental activities of daily living. Changes of instrumental activities of daily living will be assessed at the 6 weeks, 12 weeks, and 6 months.
Changes of the ADL domain of the Stroke Impact Scale | 6 months
  The ADL domain of the Stroke Impact Scale assess difficulty in performing activities of daily living. The domain score range from 10-50. A higher score indicates less difficulty in performing activities of daily living. Changes of difficulty in performing activities of daily living will be assessed at the 6 weeks, 12 weeks, and 6 months.

SECONDARY OUTCOMES:
Changes of the Fugl-Meyer Assessment | 6 months
  The Fugl-Meyer Assessment assesses ability of motor control. The total score range from 0-226. A higher score indicates better ability of motor control. Changes of ability of motor control will be assessed at the 6 weeks, 12 weeks, and 6 months.
Changes of the Mini Mental State Examination | 6 months
  The Mini Mental State Examination assesses general cognitive ability. The total score range from 0-30. A higher score indicates better general cognitive ability. Changes of general cognitive ability will be assessed at the 6 weeks, 12 weeks, and 6 months.
Changes of the Test of Visual Perceptual Skills-Third Edition | 6 months
  The Test of Visual Perceptual Skills-Third Edition assesses visual perception. The total score range from 0-112. A higher score indicates better visual perception. Changes of visual perception will be assessed at the 6 weeks, 12 weeks, and 6 months.
Changes of the Center of Epidemiological Study-Depression | 6 months
  The Center of Epidemiological Study-Depression assesses depression conditions. The total score range from 0-60. A higher score indicates more serious depression conditions. Changes of depression conditions will be assessed at the 6 weeks, 12 weeks, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Der-Sheng Han, Doctor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186